CLINICAL TRIAL: NCT02622269
Title: Patient-driven Compression in Urography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Håkan Geijer, MD, PhD, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 183781
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Urologic Diseases
Keywords: Urography; Radiation dosage; image enhancement
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient-regulated compression (Experimental): Patient-regulated compression device
  Interventions: Device: Patient-regulated compression device
- Standard compression (Active Comparator): Standard compression device
  Interventions: Device: Standard compression device

INTERVENTIONS:
Device: Patient-regulated compression device — Compression of the abdomen with a patient-regulated compression device
  Arms: Patient-regulated compression
Device: Standard compression device — Compression of the abdomen with the standard compression device
  Arms: Standard compression

SUMMARY:
Compression of the abdomen during urography with either a patient-regulated compression device or conventional compression.

Evaluation of radiation dose, image quality and patients' experiences

DETAILED DESCRIPTION:
Patients are subjected to radiation from radiographical studies. The nurse can reduce the radiation dose for the individual by using dose-reducing measures. One of these is compression. It is known that compression in urography reduces the radiation dose because the radiation has less tissue to transverse when it is compressed. By reducing patient radiation doses, the risk of harmful radiation effects is reduced. This study aims to study if a patient-regulated compression device can reduce the radiation dose as effectively as the conventional compression, regulated by the nurse.

Two compression devices are investigated in each patient, in randomized order.

Aims of the study:

1. Evaluate if the radiation doses are comparable with a patient-regulated compression device and conventional compression.
2. Evaluate image quality with the two devices.
3. Describe patients' experiences from using the two devices.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a request for a urographic study

Exclusion Criteria:

* Emergency studies,
* cannot participate actively with compression,
* contraindications to compression of the abdomen,
* pregnancy,
* inability to understand the language of the questionnaire

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Radiation dose measured as Dose-area product | Immediately
  Radiation dose for the investigated exposures, measured as Dose-area product

SECONDARY OUTCOMES:
Image quality measured with Visual Grading | Immediately
  Image quality for the investigated images, measured with Visual Grading
Patient experience (questionnaire) | Immediately after the procedure
  A questionnaire will be analysed with qualitative content analysis

CONTACTS AND LOCATIONS:
Overall Officials: Håkan Geijer, MD, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Department of Radiology, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No